CLINICAL TRIAL: NCT04596657
Title: Vitamin D3 Supplementation to Prevent Respiratory Tract Infections, Including Covid-19, in Hospital Workers: a Pragmatic Study
Brief Title: Vitamin D3 Supplementation to Prevent Respiratory Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Collaborators: Won Sook Chung Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-455
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Respiratory Tract Infections; Covid19; Flu Like Illness
MeSH Terms: conditions — Respiratory Tract Infections; COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Dietary Supplement: Vitamin D supplementation
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Vitamin D supplementation — Daily vitamin D3 supplementation (5000 IU)
  Arms: Intervention

SUMMARY:
The Cooper vitamin D3 study is a randomized study investigating whether daily vitamin D3 supplementation can prevent respiratory tract infections, influenza-like illness and covid-19 in hospital workers.

DETAILED DESCRIPTION:
Influenza-like illness and covid-19 were added to this summary because the protocol uses respiratory tract infections and influenza-like illness interchangeably. Influenza-like illness is more accurate.

Protocol amendments:

Protocol title was amended to include covid-19. Minimum age was changed from 52 to 18, expanding the sample size. Exclusion criteria re vitamin D intake was changed from >5000 to >=5000 IU.

ELIGIBILITY:
Inclusion Criteria:

* Hospital worker
* Age 18 years or older

Exclusion Criteria:

* History of hypercalcemia
* History of nephrolithiasis
* History of intolerance to vitamin D3 supplements
* Use of calcium at a dose > 600 mg/day (individuals using a dose greater than 600 mg of calcium per day will be asked to limit the amount to 600 mg unless they have been directed by their physician to be taking more than 600 mg/day of calcium. If the latter is true the potential subject will be excluded from the study.)
* Use of vitamin D at a daily dose > 5000 IU*
* Use of aluminum-containing phosphate binders in patients with renal failure
* Use of calcipotriene
* Use of digoxin
* Use of thiazide diuretics if using:

  * hydrochlorothiazide at a daily dose > 37.5 mg
  * indapamide at a daily dose > 1.25 mg
  * chlorthalidone at a daily dose > 12.5 mg
  * metolazone at a daily dose > 2.5 mg
  * methyclothiazide at a daily dose > 2.5 mg
  * chlorothiazide at a daily dose > 250 mg
  * metolazone at a daily dose > 0.5 mg
  * bendroflumethiazide at a daily dose > 2.5 mg
  * polythiazide at a daily dose > 1 mg
  * hydroflumethiazide at a daily dose > 25 mg
* Conditions that are associated with a risk of modified vitamin D metabolism
* Known allergy to wool
* Current enrollment in another study
* Life expectancy <1 month at time of screening
* Cognitive impairment precluding the ability to provide informed consent
* Pregnant or trying to become pregnant
* Employee is team member on the present study

  * If potential participants are found to be using vitamin D supplementation upon screening at a daily dose ≤5000 IU/day, they will be eligible for participation by switching to the study dose. If potential participants are taking a multiple vitamin or calcium supplement and there is less than or equal to 800 IU vitamin D in it, they can continue the multivitamin or calcium supplement along with taking the study vitamin D3. Total vitamin D cannot exceed 5,800 IU per day combined between any supplements that contain vitamin D. Use of vitamin D at a daily dose > 5000 IU at the direction of a physician will be an exclusion criterion. If a potential subject uses over-the-counter vitamin D not directed by a physician at a daily dose > 5000 IU they will be eligible to participate by switching to the lower study dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 877 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Influenza-like illness | 9 months
  Incidence of influenza-like illness

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided